CLINICAL TRIAL: NCT05591794
Title: Effects of an Eight-week Diet Versus Diet Plus Aerobic and Resistant Exercise Program on Postural Control, Musculoskeletal Disorders, Functional Capacity, and Sleep in Overweight Women: A Randomised Controlled Trial
Brief Title: Effects of Diet Versus Diet Plus Aerobic and Resistant Exercise Program in Overweight Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was halted prematurely following the departure of two researchers, resulting in insufficient research capacity to continue the study.
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant professor, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20.09.2022-78412
Record Dates: First submitted 2022-10-12; First posted 2022-10-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Exercise
Keywords: Overweight; Aerobic and resistance exercise; Postural control; Musculoskeletal disorders; Functional capacity; Sleep
MeSH Terms: conditions — Overweight; Motor Activity; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The women in the study group will be asked to walk for 30 minutes/5 days or 50 minutes/3 days a week while performing a diet program for eight weeks and aerobic and resistance exercise program 3 days a week.
  Interventions: Other: Aerobic and resistance exercises; Dietary Supplement: Diet program; Other: Regular walking program
- Control group (Active Comparator): The women in the control group will be asked to walk for 30 minutes/5 days or 50 minutes/3 days a week while performing a diet program.
  Interventions: Dietary Supplement: Diet program; Other: Regular walking program

INTERVENTIONS:
Other: Aerobic and resistance exercises — Participants in the study group will be given an aerobic exercise program on the treadmill for 8 weeks, 2 days a week, 20 minutes at a rate of 60-80% of the target heart rate. Participants will work on the treadmill for 20 minutes at 60-70% of the target heart rate for the first four weeks, and at 70-80% of the target heart rate for the last four weeks. Resistance exercises will consist of exercises that will work large muscle groups with rubber bands. According to Borg, the resistance exercises to be applied will be three sets of 10 repetitions for each movement at an RPE of 11-12 during the first four weeks, and 3 sets of 15 repetitions at the same RPE for the last four weeks, 2 times a week for 20 minutes.
  Arms: Study group
Dietary Supplement: Diet program — Initially, participants will be educated on healthy eating habits through one-on-one dietitian consultation. A personalized calorie-restricting diet will be given. According to this program, the daily energy intake of the individual will be reduced to provide 0.5-1.0 kg of body weight loss per week.
Other: Regular walking program — Regular walking will be recommended as 30 minutes/5 days or 50 minutes/3 days per week.

SUMMARY:
Adult women aged 18-50 years and overweight (preobese) with a BMI of 25-30 kg/m2 will be included in the study. Participants will participate in an eight-week diet and diet plus aerobic and resistance exercise program. Patients will be referred from the Nutrition and Diet Polyclinic of Bezmialem Vakıf University to this study, which will be conducted to investigate the effects of exercise program on postural control, musculoskeletal system disorders, functional capacity, and sleep.

DETAILED DESCRIPTION:
Subjects who accepted to participate in the study will be randomized and divided into two groups as study and control groups. A computer-based randomization program (random.org) will be used to determine the cases to be assigned to the study and control groups. 2 numbers consisting of 12 numbers will be determined by random selection from the numbers between 1 and 24. The first of these number sequences will be considered as the study group and the second as the control group. Each patient included in the study will be asked to draw one of the sealed envelopes in which the numbers 1 to 24 are written. The case will be assigned to the study or control group according to the number sequence in which the drawn number is included. While the women in the study group are expected to perform regular walking with a diet for eight weeks and a 3-day aerobic and resistance exercise program per week, the subjects in the control group will be followed up with diet and regular walking. Initially, participants will be educated on healthy eating habits through one-on-one dietitian consultation. A personalized calorie-restricting nutrition program will be given. According to this program, the daily energy intake of the individual will be reduced to provide 0.5-1.0 kg of body weight loss per week.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-29.9kg/m2
* Being between the ages of 18-50
* Agreeing to participate voluntarily in the study

Exclusion Criteria:

* Pregnancy
* Presence of systemic disease that will prevent participation in an aerobic exercise program
* Presence of conditions such as pain or surgery that will prevent participation in an aerobic exercise program
* Participating in a regular exercise program within the last 1 year

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of postural control by Biodex Balance System | Change between baseline and 8-week scores of Biodex Balance System.
  Postural control evaluation will be performed with "Biodex Balance System®" (Biodex Medical Systems, Shirley, New York, USA) which is a valid and reliable equipment. Three tests will be performed with the device: postural stability test, stability limits test, and modified clinical test of sensory integration of balance. During the evaluation, three measurements of 20 seconds, 10 seconds intervals between each measurement, will be performed in all tests. Higher control over balance is indicated by a lower score of overall, anterior/posterior, and medial/lateral stability index in the PS test. However, a higher score indicates a lower level of postural control in stability limits and modified clinical test of sensory integration of balance tests.

SECONDARY OUTCOMES:
Evaluation of musculoskeletal by Extended Nordic Musculoskeletal Questionnaire | Change between baseline and 8-week scores of Extended Nordic Musculoskeletal Questionnaire.
  The Extended Nordic Musculoskeletal Questionnaire is a reliable instrument that measures the prevalence, severity and impact of musculoskeletal symptoms.
Evaluation of functional capacity by 6 minute walk test | Change between baseline and 8-week scores of 6 Minute Walk Test.
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess functional capacity and endurance.
Evaluation of sleep quality by Pittsburgh Sleep Quality Index | Change between baseline and 8-week scores of Pittsburgh Sleep Quality Index.
  The Pittsburgh Sleep Quality Index is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Tuncer, PhD, PT, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided